CLINICAL TRIAL: NCT01190527
Title: Using FDG-PET Acquired During the Course of Radiation Therapy to Individualize Adaptive Radiation Dose Escalation in Patients With Non-Small Cell Lung Cancer
Brief Title: Using FDG-PET During Radiation Therapy in Non-Small Cell Lung Cancer
Acronym: HUM15709
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.123
Record Dates: First submitted 2010-04-01; First posted 2010-08-27 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG-PET (Other): All subjects will have the same course of treatment, the study treatment.
  Interventions: Radiation: FDG-PET

INTERVENTIONS:
Radiation: FDG-PET — This study is designed to apply functional imaging, Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) before treatment and again during treatment to see if it helps predict how well the treatment works for the cancer. The standard of care for patients with stage III unresectable NSCLC is combined chemoradiotherapy. This study will seek to determine 2 year local-regional progression free survival in patients with non-small cell lung cancer (NSCLC) when an adaptive plan is applied based on repeat PET-CT imaging during the course of radiation therapy (during RT), and investigate if there is an improvement compared to those treated with conventional radiation therapy without field and/or dose modification. The investigators hypothesize that during-RT, PET-CT-based adaptive therapy will allow them to dose escalate in the majority of patients and meet the dose limits of normal structures, thus improving local tumor control without increasing toxicity.

SUMMARY:
Successful treatment of non-small cell lung cancer with radiation therapy requires that the physicians determine exactly where the tumor is in your body, and protect your normal tissue. This study is designed to apply functional imaging, Fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) before treatment, and then again during treatment to see if the procedure helps predict how well the treatment works for your cancer and how well your lung functions during treatment. FDG-PET is a modern technology that uses small amounts of a radioactive glucose (FDG) to make images of your whole body and areas of active cancer. A Computerized Tomography (CT) will also be performed along with both of these procedures to help the researchers see clearly where your cancer or your healthy lung is located. The study will help the investigator determine whether an adaptive plan that is applied based on repeat PET-CT imaging during the course of radiation therapy (during RT), can show if there is an improvement in treatment outcome compared to those treated with standard radiation therapy. This adaptive plan may allow your doctor to escalate the dose per treatment and the total dose of your treatment based on the risk of damage to your healthy lung tissue. While increasing the radiation dose, but limiting the toxicity to normal lung tissue, the researchers hope to improve your tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid and pathologically proven non-small cell lung cancer. If pathology not definitive, the patient needs to have a clinically diagnosed non-small cell lung cancer, which is also FDG-avid.
* Patients must be 18 years of age or older.
* Patients must have Karnofsky performance score > 60.
* Patients must have clinical AJCC (American Joint Committee on Cancer) Stage I-IIIB, with unresectable or inoperable disease.
* Patients must have no evidence of a malignant pleural or pericardial effusion
* Patients must have hemoglobin > 10 gm/dl. Transfusions or medications may be used to achieve this criterion.
* Patients must have reasonable organ and marrow functions as defined below if chemotherapy is considered:

  * WBC (White Blood Cell) > 3,000/mm3.
  * absolute neutrophil count ≥ 1,500/mm3.
  * platelets > 100,000/mm3
  * total bilirubin ≤ 3.0 mg/dl.
  * AST ( Aspartate Aminotransferase or SGOT) and ALT (Alanine Transaminase or SGPT) < 4 X institutional upper limit of normal.
  * creatinine ≤ 2.0 mg/dl.
* Patients must not have serious intercurrent diseases per the judgment of the treating physician.
* Patient must be willing to use effective contraception if female with reproductive capability.
* Patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients with any component of small cell lung carcinoma are excluded from this study.
* Prior radiotherapy to the thorax such that composite radiation would significantly overdose critical structures, either per estimation of the treating radiation oncologist or defined by failure to meet normal tissue tolerance constraints.
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects.
* Prisoners are excluded for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2014-07 (Actual); Study Completion 2015-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Kong FM, Ten Haken RK, Schipper M, Frey KA, Hayman J, Gross M, Ramnath N, Hassan KA, Matuszak M, Ritter T, Bi N, Wang W, Orringer M, Cease KB, Lawrence TS, Kalemkerian GP. Effect of Midtreatment PET/CT-Adapted Radiation Therapy With Concurrent Chemotherapy in Patients With Locally Advanced Non-Small-Cell Lung Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2017 Oct 1;3(10):1358-1365. doi: 10.1001/jamaoncol.2017.0982. PMID 28570742

RESULTS

PARTICIPANT FLOW:
Groups:
- Adaptive Radiation: Conformal radiotherapy (RT) was given in 30 daily fractions. RT dose was individualized to a fixed risk of lung toxicity and adaptively escalated to the residual tumor on mid-tx FDG-PET up to a total physical dose of 86 Gy.
Period: Overall Study
Arm/Group | Adaptive Radiation
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adaptive Radiation
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Rate of Overall Local-Regional Tumor Control Using FGD-PET-CT During Radiation Therapy(RT)
Description: Use FGD-PET-CT based adaptive radiation to deliver a higher total dose to the active tumor to determine if it will improve the local-regional tumor control and progression-free survival in patients, without increasing the normal tissue complication probability (NTCP) of the lung.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Adaptive Radiation
Number analyzed (Participants) | 42
percentage of patients | 68 [47 to 82]

2. Secondary Outcome: Number of Patients That Were Able to Receive Dose Escalation
Description: The number of patients for which dose escalation was possible will be reported.
Time Frame: 2 Years
Measure: Number; unit: participants
Arm/Group | Adaptive Radiation
Number analyzed (Participants) | 42
participants | 42

3. Secondary Outcome: Percentage of Patients Alive at 2 Years
Description: Overall survival of all patients will be estimated
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Adaptive Radiation
Number analyzed (Participants) | 42
percentage of patients | 51 [34 to 65]

4. Secondary Outcome: The Number of Participants That Experience Lung Toxicity and Esophagitis
Description: The number of participants that experience RT (radiation therapy) induced lung toxicity, and grade 2 or greater (symptomatic) esophagitis, will be recorded.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Adaptive Radiation
Number analyzed (Participants) | 42
participants
  RT-induced lung toxicity | 8
  esophagitis (grade 2 or greater) | 13

ADVERSE EVENTS:
Arm/Group | Adaptive Radiation
Serious Adverse Events (participants affected / at risk) | 29/42
Other Adverse Events (participants affected / at risk) | 30/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Radiation (N=42)
Allergic reaction (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Asystole (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Bladder infection (Renal and urinary disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cardiac pain (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constitutional Symptoms - Other (Specify) (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Esophagitis (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu-like syndrome (Infections and infestations) | 1 (1)
Gait abnormal (Nervous system disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage - Other (Specify) (Vascular disorders) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Cardiac disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Infection - Other (Specify) (Infections and infestations) | 1 (2)
Infection, Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Infection, Prostate (Reproductive system and breast disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Laryngeal edema (Gastrointestinal disorders) | 1 (2)
Left ventricular diastolic dysfunction (Cardiac disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutrophils (Blood and lymphatic system disorders) | 1 (1)
PTT (Investigations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary - Other(specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Sudden death (General disorders) | 3 (3)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Voice alteration (Gastrointestinal disorders) | 1 (1)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adaptive Radiation (N=42)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (7)
Anxiety (Psychiatric disorders) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cardiac General - Other (Specify) (Cardiac disorders) | 3 (5)
Chest pain (Cardiac disorders) | 5 (7)
Chest wall pain (Cardiac disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (19)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 3 (6)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 16 (29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (37)
Edema limbs (General disorders) | 3 (4)
Esophageal pain (Gastrointestinal disorders) | 4 (7)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 17 (32)
Fever (General disorders) | 4 (7)
Headache (Nervous system disorders) | 5 (7)
Hemoglobin (Blood and lymphatic system disorders) | 9 (19)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (38)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Hyponatremia (Metabolism and nutrition disorders) | 6 (9)
Hypotension (Cardiac disorders) | 3 (5)
Leukocytes (Blood and lymphatic system disorders) | 9 (20)
Lymphopenia (Blood and lymphatic system disorders) | 17 (46)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (11)
Neutrophils (Blood and lymphatic system disorders) | 11 (13)
Pericardial effusion (Cardiac disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Pharyngolaryngeal pain (Gastrointestinal disorders) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Pulmonary - Other(specify) (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 (20)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (5)
Weight loss (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes